CLINICAL TRIAL: NCT04643964
Title: Building Mental Health Resilience in the COVID-19 Pandemic.
Brief Title: Brief Video Interventions for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Daniel R. Strunk, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020B0326
Record Dates: First submitted 2020-11-12; First posted 2020-11-25 (Actual); Results first posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Depressive Symptoms
Keywords: Depression; Video intervention; Cognitive behavioral skills
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three conditions: (1) a brief intervention focused on one domain of coping skills (the entrée condition), (2) a brief intervention focused on three domains of coping skills (the sampler condition), or (3) a no-intervention control condition. If participants are randomly assigned to the first condition, they will be further randomized into one of three brief interventions: (1) a focus on cognitive coping skills, (2) a focus on behavioral coping skills, or (3) a focus on interpersonal coping skills. The sampler condition will involve limited coverage of each of these same three types of skills.
Masking Description: Participants are told they may or may not be asked to watch videos and fill out worksheets. More detailed descriptions of the interventions being tested are not provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Entrée: Cognitive Skills (Experimental)
  Interventions: Behavioral: Entrée: Cognitive skills
- Entrée: Behavioral Skills (Experimental)
  Interventions: Behavioral: Entrée: Behavioral skills
- Entrée: Interpersonal Skills (Experimental)
  Interventions: Behavioral: Entrée: Interpersonal skills
- Sampler Skills (Experimental)
  Interventions: Behavioral: Sampler skills
- Control (No Intervention): Participants are not given videos to watch until their involvement in the study ends.

INTERVENTIONS:
Behavioral: Entrée: Cognitive skills — In this condition, participants view a video-based intervention covering cognitive emotion regulation skills. This intervention asks participants to respond to questions and practice identifying and evaluating their own thoughts using an intervention worksheet. One week after the intervention, participants are asked to upload a worksheet showing their efforts to use the intervention skills.
  Arms: Entrée: Cognitive Skills
Behavioral: Entrée: Behavioral skills — In this condition, participants view a video-based intervention covering behavioral emotion regulation skills. This intervention asks participants to respond to questions and practice scheduling activities that might give them a sense of pleasure or accomplishment using an intervention worksheet. One week after the intervention, participants are asked to upload a worksheet showing their efforts to schedule and engage in behaviors in line with the intervention skills.
  Arms: Entrée: Behavioral Skills
Behavioral: Entrée: Interpersonal skills — In this condition, participants view a video-based intervention covering interpersonal emotion regulation skills. This intervention asks participants to respond to questions and practice communicating effectively using an intervention worksheet. One week after the intervention, participants are asked to upload a worksheet showing their efforts to use the intervention skills.
  Arms: Entrée: Interpersonal Skills
Behavioral: Sampler skills — In this condition, participants view a video-based intervention covering three emotion regulation skills: cognitive, behavioral, and interpersonal skills. This intervention asks participants to respond to questions and practice using skills using intervention worksheets. One week after the intervention, participants are asked to upload a worksheet showing their efforts to use the intervention skills.
  Arms: Sampler Skills

SUMMARY:
In this study, we test brief video interventions for those with elevated depressive symptoms. We randomize participants to one of three conditions. (1) An entrée condition involving in-depth coverage a set of cognitive behavioral therapy (CBT) skills. (2) A sampler condition which introduces three sets of CBT skills. (3) A control condition involving no skills. Among those in the entrée condition, participants are further randomized to one of three CBT skills. We plan on two sets of primary comparisons. First, we will compare the effects of each form of video intervention (i.e., entrée and sampler) to the control condition. Second, we will compare the entrée and sampler conditions. We will recruit participants from Amazon's Mechanical Turk program (MTurk). In the intervention conditions, participants will be asked to watch several videos and practice skills using worksheets. They will also be asked to practice skills introduced in the videos in the week following the intervention. In the control condition, participants will not watch videos. One week after the intervention, all participants will respond to a follow-up assessment.

DETAILED DESCRIPTION:
Access to the study will be provided via the MTurk website. Study measures and interventions will be provided via Qualtrics. To determine eligibility, participants will be asked to fill out a pre-screening measure of depressive symptoms, the Personal Health Questionnaire-9 (PHQ-9). Those who score 10 or higher will be eligible. After consenting to participate, participants will fill out baseline measures, be randomly assigned to a condition, participate in any condition related procedures, and then respond to a follow-up assessment one week later.

Each brief intervention consists of watching a series of videos. After each video, participants in the intervention conditions will be prompted to answer a series of questions to practice the skills explained in the videos. For the entrée and sampler conditions, watching all videos and filling out any worksheets that are part of the initial intervention is expected to take approximately 30 minutes.

Participants in the entrée and sampler conditions will be asked to work on a coping skills worksheet over the next seven days (estimated to involve about 10 minutes of work). Participants will receive an email seven days after participating in the brief intervention, asking them to take part in the following portion of the study. Before beginning the follow-up activity, participants in the intervention conditions will be asked to upload the coping skills worksheet they worked on. All participants will be asked to respond to follow-up assessment measures at this point.

ELIGIBILITY:
Inclusion Criteria:

* Score above 10 on the Patient Health Questionnaire-9
* Are 18 years of age or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 655 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2021-06-05 (Actual); Study Completion 2021-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Strunk, Ph.D., Principal Investigator — Ohio State University
Locations (1):
- Department of Psychology, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Results will be posted to clinicaltrials.gov within one year after completion of the final participant's participation in the clinical trial. Following initial publication, deidentified individual participant data (IPD) that underlie results in the primary outcome data reported will be available on reasonable request for 5 years after study completion.
Time Frame: IPD will be available upon reasonable request within one year of primary outcome manuscript being published.
Access Criteria: Proposals should be directed to Daniel R. Strunk at strunk.20@osu.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 951 participants were eligible. 272 participants discontinued before randomization, 6 participants did not provide sufficient identification to invite them to Time 2 of the study, and 18 participants attempted to complete Time 1 multiple times.
Period: Overall Study
Arm/Group | Entrée: Cognitive Skills | Entrée: Behavioral Skills | Entrée: Interpersonal Skills | Sampler Skills | Control
Started | 86 | 90 | 89 | 258 | 132
Completed | 30 | 23 | 33 | 115 | 73
Not Completed | 56 | 67 | 56 | 143 | 59
Not completed — Lost to Follow-up | 55 | 59 | 54 | 129 | 48
Not completed — Failed attention check | 1 | 8 | 2 | 14 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Entrée: Cognitive Skills | Entrée: Behavioral Skills | Entrée: Interpersonal Skills | Sampler Skills | Control | Total
Number analyzed (Participants) | 86 | 90 | 89 | 258 | 132 | 655
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Number differs because some participants did not enter their age.
  years
    number analyzed (Participants) | 86 | 88 | 89 | 257 | 132 | 652
    (all) | 36.15 (10.29) | 34.95 (9.67) | 37.07 (11.40) | 35.50 (10.63) | 36.48 (11.63) | 35.93 (10.77)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 49 | 49 | 50 | 140 | 75 | 363
  Male | 35 | 37 | 36 | 110 | 49 | 267
  Another gender | 2 | 4 | 3 | 8 | 7 | 24
  Did not give | 0 | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaska Native | 0 | 1 | 1 | 2 | 0 | 4
  Asian | 6 | 7 | 4 | 21 | 6 | 44
  Black | 13 | 19 | 16 | 30 | 17 | 95
  Hispanic/Latino | 5 | 8 | 7 | 15 | 6 | 41
  Middle Eastern/North African | 1 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian/Pacific Islander | 1 | 0 | 0 | 1 | 1 | 3
  White | 50 | 48 | 56 | 172 | 100 | 426
  Other/multi-racial | 10 | 7 | 5 | 16 | 2 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in the Quick Inventory of Depressive Symptoms-Self Report (QIDS-SR)
Description: The Quick Inventory of Depressive Symptoms-Self Report is a 16-item self-report scale that measures depressive symptom severity. Scores range from 0 to 27, with higher scores indicating greater depressive symptoms.
Time Frame: Baseline, 1-2 weeks after baseline
Population: Number differs because: (1) some participants did not enter information in to complete the measure, and (2) some participants did not move on to Time 2.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Entrée: Cognitive Skills | Entrée: Behavioral Skills | Entrée: Interpersonal Skills | Sampler Skills | Control
Number analyzed (Participants) | 86 | 90 | 89 | 258 | 132
units on a scale
  Time 1, Baseline: number analyzed (Participants) | 86 | 89 | 89 | 258 | 131
  Time 1, Baseline | 13.67 (3.90) | 14.09 (4.67) | 14.29 (4.15) | 13.79 (4.38) | 14.03 (4.38)
  Time 2, 1-2 weeks after baseline: number analyzed (Participants) | 30 | 22 | 33 | 116 | 77
  Time 2, 1-2 weeks after baseline | 13.00 (4.32) | 11.91 (5.61) | 12.94 (4.44) | 11.47 (4.72) | 12.60 (5.36)
Statistical Analysis 1: Comparison: Entrée: Cognitive Skills vs Entrée: Behavioral Skills vs Entrée: Interpersonal Skills vs Sampler Skills vs Control; In this model, the condition included the following levels: entrée, sampler, and control. No covariates were included; Test type: Superiority; p = .54, ANCOVA

2. Secondary Outcome: Change in the Ways of Responding Questionnaire (WOR)
Description: The Ways of Responding Questionnaire is a measure of compensatory skills taught in CBT for depression. Participants respond to 6 hypothetical stressful situations in which their initial thoughts regarding the event are given. Quality scores range from 0 to 6, with higher scores indicating greater CBT skills.
Time Frame: Baseline, 1-2 weeks after baseline
Population: Number differs because: (1) some participants did not enter information in to complete the measure, (2) some participants did not move on to Time 2, and (3) some participants entered in data that was not possible to code (e.g., "N/A").
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Entrée: Cognitive Skills | Entrée: Behavioral Skills | Entrée: Interpersonal Skills | Sampler Skills | Control
Number analyzed (Participants) | 86 | 90 | 89 | 258 | 132
units on a scale
  Time 1, Baseline: number analyzed (Participants) | 41 | 39 | 44 | 137 | 88
  Time 1, Baseline | 3.58 (.92) | 3.70 (.95) | 3.71 (.75) | 3.70 (.87) | 3.7 (.88)
  Time 2, 1-2 weeks after baseline: number analyzed (Participants) | 21 | 15 | 26 | 83 | 53
  Time 2, 1-2 weeks after baseline | 3.88 (.97) | 4.08 (.94) | 3.87 (.75) | 4.02 (1.01) | 3.96 (1.02)
Statistical Analysis 1: Comparison: Entrée: Cognitive Skills vs Entrée: Behavioral Skills vs Entrée: Interpersonal Skills vs Sampler Skills vs Control; In this model, the condition included the following levels: entrée, sampler, and control. There was one covariate in this model: QIDS at Time 1; Test type: Superiority; p = .92, ANCOVA

3. Secondary Outcome: Change in the Styles of Emotion Response Questionnaire (SERQ)
Description: The Styles of Emotion Response Questionnaire is a 36-item self-report scale that measures the extent to which respondents endorse four different domains of coping skills: cognitive, behavioral, interpersonal, and mindfulness. For each item, participants are asked how often they use the strategy and how much feeling upset negatively impacts the use of this strategy. Scores from the first three skills are secondary outcomes. Scores range from 72-360, with higher scores indicating greater coping skill use.
  For the purpose of this study, we used the Cognitive, Behavioral, and Interpersonal scales. Scores in each subscale range from 18-90, with higher scores indicating greater coping skill use in that domain.
Time Frame: Baseline, 1-2 weeks after baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Entrée: Cognitive Skills | Entrée: Behavioral Skills | Entrée: Interpersonal Skills | Sampler Skills | Control
Number analyzed (Participants) | 86 | 90 | 89 | 258 | 132
units on a scale
  Cognitive Subscale: Time 1, Baseline: number analyzed (Participants) | 84 | 89 | 87 | 251 | 129
  Cognitive Subscale: Time 1, Baseline | 33.45 (6.80) | 32.85 (6.50) | 33.31 (5.31) | 32.69 (7.56) | 32.57 (7.43)
  Cognitive Subscale: Time 2, 1-2 weeks after baseline: number analyzed (Participants) | 29 | 23 | 33 | 116 | 76
  Cognitive Subscale: Time 2, 1-2 weeks after baseline | 33.41 (6.96) | 32.61 (6.62) | 34.12 (5.99) | 34.04 (7.56) | 33.31 (7.53)
  Behavioral Subscale: Time 1, Baseline: number analyzed (Participants) | 83 | 86 | 88 | 253 | 127
  Behavioral Subscale: Time 1, Baseline | 33.31 (8.09) | 31.36 (7.86) | 32.44 (6.02) | 31.84 (8.35) | 31.32 (8.06)
  Behavioral Subscale: Time 2, 1-2 weeks after baseline: number analyzed (Participants) | 29 | 23 | 33 | 116 | 76
  Behavioral Subscale: Time 2, 1-2 weeks after baseline | 35.17 (6.85) | 34.13 (6.88) | 32.88 (6.91) | 33.22 (8.18) | 32.73 (8.14)
  Interpersonal Subscale: Time 1, Baseline: number analyzed (Participants) | 83 | 89 | 88 | 253 | 128
  Interpersonal Subscale: Time 1, Baseline | 32.11 (7.50) | 30.38 (8.31) | 30.75 (6.73) | 30.53 (8.37) | 30.88 (8.43)
  Interpersonal Subscale: Time 2, 1-2 weeks after baseline: number analyzed (Participants) | 29 | 23 | 33 | 116 | 76
  Interpersonal Subscale: Time 2, 1-2 weeks after baseline | 33.38 (6.75) | 31.43 (7.44) | 31.15 (6.49) | 31.16 (8.44) | 31.16 (8.34)
Statistical Analysis 1: Comparison: Entrée: Cognitive Skills vs Entrée: Behavioral Skills vs Entrée: Interpersonal Skills vs Sampler Skills vs Control; In this model, the condition included the following levels: entrée, sampler, and control. There were three covariates in this model: QIDS at Time 1, gender, and COVID interference; Test type: Superiority; p = .37, ANCOVA

4. Secondary Outcome: Change in the University of California, Los Angeles (UCLA) Loneliness Scale, Version 3
Description: The University of California, Los Angeles (UCLA) Loneliness Scale, Version 3 is a 20-item self-report scale that measures subjective feelings of loneliness and isolation. Scores range from 20-80, with higher scores indicating greater subjective experience of loneliness.
Time Frame: Baseline, 1-2 weeks after baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Entrée: Cognitive Skills | Entrée: Behavioral Skills | Entrée: Interpersonal Skills | Sampler Skills | Control
Number analyzed (Participants) | 86 | 90 | 89 | 258 | 132
units on a scale
  Time 1, Baseline: number analyzed (Participants) | 82 | 87 | 88 | 251 | 127
  Time 1, Baseline | 53.87 (9.16) | 55.80 (9.25) | 54.70 (9.22) | 53.97 (9.53) | 54.66 (10.10)
  Time 2, 1-2 weeks after baseline: number analyzed (Participants) | 30 | 23 | 33 | 116 | 77
  Time 2, 1-2 weeks after baseline | 52.59 (10.54) | 54.57 (10.76) | 56.83 (8.16) | 53.20 (10.40) | 54.20 (10.80)
Statistical Analysis 1: Comparison: Entrée: Cognitive Skills vs Entrée: Behavioral Skills vs Entrée: Interpersonal Skills vs Sampler Skills vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .87, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse event data were not collected.
Description: Adverse event data were not collected.
Arm/Group | Entrée: Cognitive Skills | Entrée: Behavioral Skills | Entrée: Interpersonal Skills | Sampler Skills | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT04643964/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/64/NCT04643964/SAP_001.pdf